CLINICAL TRIAL: NCT00988806
Title: Double-blind Randomized Placebo-controlled Study to Evaluate the Efficacy and Safety of Intermittent, Long-term Administration of Levosimendan in Patients With Advanced Heart Failure
Brief Title: Long-Term Intermittent Administration of Levosimendan in Patients With Advanced Heart Failure
Acronym: LAICA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Principal Investigator, Martín J García González, Consultant MD, PhD, Hospital Universitario de Canarias
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAICA Study 2009; EudraCT 2009-011441-11
Record Dates: First submitted 2009-09-29; First posted 2009-10-02 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Advanced Heart Failure
Keywords: Advanced heart failure; Levosimendan; Intermittent long-term infusions
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levosimendan (Active Comparator): infusion of levosimendan at doses of 0.1 mcg / kg / min for 24 hours.
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): infusion of placebo for 24 hours.
  Interventions: Drug: Levosimendan; Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — Patients included in the intervention group receive optimal drug therapy for heart failure symptoms and also infusion of levosimendan at doses of 0.1 mcg / kg / min for 24 hours every 30 days.
  Failure to reach an appropriate level of heart failure compensation before the deadline of 30 days for the next study drug administration or placebo, the administration of them will be every 15 days. Thereafter, failure to reach an appropriate level of heart failure compensation for patients or worsen after two consecutive infusions of study drug or placebo every 15 days, proceed to open the code patient randomization and and apply the most appropriate treatment.
Drug: Placebo — Patients included in the placebo group receive optimal drug therapy for heart failure and also infusion of placebo at the same infusion rate as levosimendan doses of 0.1 mcg / kg / min for 24 hours every 30 days.
  Failure to reach an appropriate level of heart failure compensation before the deadline of 30 days for the next study drug administration or placebo, the administration of them will be every 15 days. Thereafter, failure to reach an appropriate level of heart failure compensation for patients or worsen after two consecutive infusions of study drug or placebo every 15 days, proceed to open the code patient randomization and and apply the most appropriate treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the treatment strategy of long-term intermittent every 30 days, continuous intravenous infusion for 24 hours of Levosimendan, associated to optimal contemporary treatment for advanced heart failure reduce the incidence of admission for heart failure worsening at 12 months follow up, compared with the strategy based solely in the optimal contemporary treatment for advanced heart failure.

DETAILED DESCRIPTION:
Aims: To evaluate the efficacy and safety of long-term, intermittent intravenous administration for 24 hours of Levosimendan for the treatment of advanced heart failure. Main end-point: incidence of admission due to decompensation, defined as first admission to emergency services or hospitalization more than 12 hours due to heart failure worsening.

Secondary end-points: major cardiac events, serious adverse events, change in NYHA scale at baseline, 30 days, 6 and 12 months; effects on inflammatory and neurohormonal activation in heart failure, identify factors associated with better survival of patients, quality of life, cost-effectiveness of treatment.

Study Design: Prospective, randomized, double-blind placebo controlled trial.

Scope of the study: patients with advanced heart failure.

Study Subjects: Patients over 18 years old with advanced HF of any etiology, with at least one admission for acute decompensation treated or treatable with Levosimendan within 6 months prior to randomization.

Interventions: a 24-hour infusion every 30 days of Levosimendan or placebo in addition to optimal pharmacological treatment for HF during 12 months.

Determinations: clinical monitoring, protocol-specified analytical determinations, echocardiographic assessment, invasive hemodynamic assessment, functional assessment by 6 min walk test in corridor, quality of life assessment at baseline, after 30 days, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Severe symptoms of heart failure with dyspnea and/or fatigue at rest or minimal effort (functional class III and IV of NYHA)
* Episodes of fluid retention (pulmonary or systemic venous congestion, peripheral edema) and/or low cardiac output at rest (peripheral hypoperfusion)
* objective evidence of severe cardiac dysfunction determined by the presence of at least one of the following:
* Left ventricular ejection fraction </= 30%
* A severe impairment of cardiac function by echocardiography with Doppler transmitral flow pattern pseudonormal or restrictive.
* A left ventricular filling pressure elevated (PCP> 16 mmHg and / or DBP average> 12 mm Hg for pulmonary artery catheterization)
* Levels of BNP or NT-proBNP higher in the absence of noncardiac causes for this.
* Severe impairment of functional capacity as evidenced by one of the following:
* Inability to exercise
* A distance <300 m or less in women and / or patients >/= 75 years in the 6-minute walk test
* A test of myocardial oxygen consumption <12-14 ml / kg / min.
* >/= 1 prior history of HF hospitalization in the previous 6 months
* Presence of all the above criteria despite attempts to optimize therapy including diuretics, inhibitors of the renin-angiotensin-aldosterone system and beta-blockers, unless these drugs were not tolerated or were contraindicated, and cardiac resynchronization therapy when indicated.
* consent to participate in the study.

Exclusion Criteria:

* Levosimendan allergy or hypersensitivity.
* Severe renal impairment (creatinine clearance <30 ml / min).
* Severe liver impairment.
* History of autoimmune disease.
* Pregnancy.
* Women of childbearing age not using adequate contraception (hormonal, IUD, barrier + spermicide)
* Heart disease with significant obstructions to ventricular filling or emptying.
* Severe hypotension (Systolic < 90 mmHg).
* Tachycardia > 120 bpm or a history of torsion point type ventricular tachycardia.
* Severe concomitant disease with decreased short-term prognosis.
* Inability to give informed consent.
* Participation in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of admission for heart failure worsening in patients with advanced heart failure, defined as first admission to emergency services or hospitalization more than 12 hours due to a heart failure worsening. | one year

SECONDARY OUTCOMES:
Time from randomization until first hospitalization for heart failure worsening. All-cause mortality. Major cardiac events. Serious adverse events. Changes in NYHA scale and quality of life of patients. To analyze the cost-effectiveness of treatment. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Martín J García González, MD, PhD, Principal Investigator — Hospital Universitario de Canarias. La Laguna. Tenerife. Spain
Locations (1):
- Department of Cardiology. Hospital Universitario de Canarias, San Cristóbal de La Laguna, S.C. de Tenerife, Spain

REFERENCES:
- [Background] Garcia-Gonzalez MJ, de Mora-Martin M, Lopez-Fernandez S, Lopez-Diaz J, Martinez-Selles M, Romero-Garcia J, Cordero M, Lara-Padron A, Marrero-Rodriguez F, del Mar Garcia-Saiz M, Aldea-Perona A; LAICA study investigators. Rationale and design of a randomized, double-blind, placebo controlled multicenter trial to study efficacy, security, and long term effects of intermittent repeated levosimendan administration in patients with advanced heart failure: LAICA study. Cardiovasc Drugs Ther. 2013 Dec;27(6):573-9. doi: 10.1007/s10557-013-6476-7. PMID 23887741